

University Hospitals of Leicester NHS

National Institute for Health Research Leicester Respiratory Biomedical Research Unit

> Glenfield Hospital Groby Road Leicester LE3 9QP

Telephone: 07414638380 Email: t.ward@lboro.ac.uk

www.leicsrespiratorybru.nihr.ac.uk

IRAS ID: 243125

Date and version number: Version 1.2,

13.07.2018

Participant Identification Number:

## **CONSENT FORM (COPD)**

Title of Project: Personalised exercise training in COPD – comprehensive phenotyping of exercise training response Name of Researcher: Please initial box 1. I confirm that I have read the information sheet dated 13.07.18 v1.2 for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. 3. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from Loughborough University, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. 4. I agree to identifiable information being transferred securely to Loughborough University 5. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers. 6. I understand that my anonymised data will be aggregated for analysis and publication of the results of the study and I will be given a summary of these results 7. I agree to my General Practitioner being informed of my participation in the study. 8. I agree to take part in the above study. Name of Participant Date Signature Name of Person taking consent Date Signature